CLINICAL TRIAL: NCT01433029
Title: Objective Assessment of Technical Skills in Cardiothoracic Surgery
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0595
Record Dates: First submitted 2011-09-08; First posted 2011-09-13 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Other Surgical Procedures
Keywords: Surgical Procedure; Assessment; Cardiothoracic Surgery; Coronary artery bypass; CAB; Video recordings; Global rating scale; GRS; Cardiothoracic surgeon; Surgical trainees

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Conventional Rater (CR): CR Group receives conventional training from PI about how to rate coronary artery bypass (CAB) videos.
  Interventions: Other: Surgical Video Assessments
- Video Rater (VR): VR Group receives conventional training from PI about how to rate CAB videos, along with a video rater training manual.
  Interventions: Other: Surgical Video Assessments
- CAB Recording: CAB recording of performance cardiothoracic surgeon or surgical trainee in 1st, 2nd, or 3rd year of training.
  Interventions: Other: Video Recording of CAB

INTERVENTIONS:
Other: Surgical Video Assessments — Rate performance of the surgeon/trainee in each CAB video performance (5 recorded procedures) using two rating scales, a checklist and the Global Rating Scale. Up to 38 different recorded procedures rated while on the study, each procedure lasting about 15 minutes.
  Groups: Conventional Rater (CR); Video Rater (VR)
Other: Video Recording of CAB — Each video begins when dissection of a coronary artery has begun and ends when all manipulation of anastomosis is complete. At least 6 separate anastomoses will be recorded, or at least 2-3 procedures. A ProXennon Surgical Headlight Camera System (a small camera that is mounted in place directly over a high-intensity light that is worn on the head) records the performance of the coronary artery bypass (CAB) procedures.
  Groups: CAB Recording

SUMMARY:
The goal of this research study is to develop a method of rating videos of CAB procedures that will produce a reliable assessment of a cardiothoracic surgical trainee's technical proficiency. In addition, researchers also want to learn if using a video manual to train raters can help improve rater reliability.

DETAILED DESCRIPTION:
Cardiothoracic Surgeon:

If you agree to take part in this study, you will receive a DVD containing multiple videos of different surgeons or surgical trainees performing CAB procedures. You will be trained by the Principal Investigator (PI) on how you should rate the performance of each surgeon/trainee. You will be randomly assigned to 1 of 2 groups:

* If you are in the Conventional Rater (CR) Group, you will receive conventional training from the PI about how to rate the videos.
* If you are in the Video Rater (VR) Group, you will receive conventional training from the PI about how to rate the videos. You will also receive a video rater training manual.

You will receive up to 38 different recorded procedures while you are on study. Each procedure should last about 15 minutes. You will record the identification code that appears at the beginning of each video, and the date and time that you viewed each video. You will watch each video and then rate the performance of the surgeon/trainee using a checklist and a Global Rating Scale. These rating documents will be given to you on a thumb drive that you will either fill out on your computer or print out and fill in by hand. You will be given more detailed instructions on how to fill out the checklist and rating scales by the Principal Investigator (PI).

Your identity will be coded and blinded throughout the study. No identifying information will be directly linked to your responses. Only the video identification numbers and your code number will be used to identify the assessment data. The code key will be stored in a separate computer or thumb drive.

Length of Study:

You will have 1 month to view and rate all videos. You will be contacted 1 time each week by the PI to monitor your progress.

After you have watched and rated all the videos, you will return the videos, your responses (either on the thumb drive or on printed hard-copies), and the video rater training manual (if you are in the VR group) in a pre-paid mailer.

Up to 20 raters may take part in this study.

Cardiothoracic Surgical Trainee:

If you agree to take part in this study, you will fill out a form that asks about your surgical experience. It will also ask about your age, sex, and initials, but these fields are optional.

You will then use the ProXennon Surgical Headlight Camera System (a small camera that is mounted in place directly over a high-intensity light that you wear on your head) to record yourself performing CAB procedures. The main principal investigator (PI) will be present when the system is being used to make sure that it is set up properly and to collect the videos when the procedures are complete. No audio will be recorded. Each video will begin when the dissection of a coronary artery has begun and will end when all manipulation of the anastomosis is complete. You will record at least 6 separate anastomoses, or at least 2-3 procedures.

The time taken to set-up the recording equipment will be documented by the PI for each procedure. After each procedure, a questionnaire will be completed by the intra-operative personnel (nurses, anesthesiologist, perfusionist, operative surgeon, assistant surgeon) that contains questions about any interference from the recording equipment. Neither you nor the intra-operative personnel will be identified in this questionnaire.

The videos will be given a code number. The code key will be kept separately from the video recordings. No identifying information will be directly linked to your videos. Only the researcher in charge will have access to the code key. This is so the researcher will be able to link the videos to the form you filled out at the beginning of the study describing your surgical experience. All data will be presented in aggregate to protect participant identity.

Length of Study:

Your participation in this study will be over after you have submitted your last recording

This is an investigational study. The ProXennon Surgical Headlight Camera System is an approved, standard method of recording CAB procedures.

Up to 22 trainees and up to 8 experienced surgeons may take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The trainee must be a cardiothoracic surgical trainee in their 1st, 2nd, or 3rd year of training and must be currently enrolled at any of the following institutions: U.T. Health Science Center in Houston, The Texas Heart Institute/Baylor College of Medicine, U.T. San Antonio, U. T. Southwestern, U.T. M.D. Anderson Cancer Center, and The Methodist Hospital.
2. The trainee must provide an informed consent to participate.
3. The experience faculty must be a cardiothoracic surgeon who regularly performs CAB procedures and has at least 10 years of post-training experience.
4. The experienced faculty is currently operating at the same institutions listed in inclusion criterion 1.
5. The experienced faculty must provide written informed consent to participate.
6. The faculty rater must be a cardiothoracic surgeon who regularly performs CAB procedures, is practicing in an Adult Cardiothoracic Graduate Medical Evaluation (ACGME) approved CTS training program, and has practiced at least 5 years after certification by the American Board of Thoracic Surgery (ABTS). There is no restriction on geographic location.
7. The expert CAB surgeon for Consensus Building must be a cardiothoracic surgeon who regularly performs CAB procedures, is practicing in an ACGME approved CTS training program, and has practiced at least 10 years after certification by the ABTS. There is no restriction on geographic location.

Exclusion Criteria:

N/A

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiothoracic surgical trainee in their 1st, 2nd, or 3rd year of training. Experienced faculty are cardiothoracic surgeons who regularly perform coronary artery bypass (CAB) procedures and have at least 10 years of post-training experience.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2017-01-22 (Actual); Study Completion 2017-01-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of Video Recordings of Cardiothoracic Surgery (CTS) Procedures | 1 month for rating
  Assessing 5 recorded procedures with qualified raters using two rating scales; a checklist developed using a consensus building project and a global rating scale (GRS) adapted from an established surgical assessment tool. The GRS uses a 5 point scale and behavioral anchors are provided for 1, 3, and 5 (a score of 1 equals a novice, 3 equals a competent surgeon, and 5 equals an expert). Raters have 1 month to view videos.

CONTACTS AND LOCATIONS:
Overall Officials: Ara Vaporciyan, MD,BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - The University of Texas Southwestern Medical Center in Dallas, Dallas, Texas
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org